CLINICAL TRIAL: NCT03980665
Title: The Effect of Arsenic Trioxide on Eliminating HIV-1 Reservoir Combined With cART
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Guangzhou Institutes of Biomedicine and Health Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Linghua LI, Vice Chief physician, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170812V1
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS
Keywords: Arsenic Trioxide; cART; HIV-1 reservoir; functional cure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Arsenic Trioxide

STUDY DESIGN:
Intervention Model Description: The control arm includes HIV-infected patients with the therapy of Antiretroviral drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arsenic trioxide combined with cART (Experimental): Receiving intravenous arsenic trioxide, 0.16mg/kg/day, no more than 10 mg per-day , two to four weeks, combined with continuous cART after attaining plasma HIV-1 suppression (plasma HIV RNA <50 cp/ml) and CD4+ cell count more than 350 cells/ul over 1 year by cART, without active HCV or HBV infection or opportunistic infections.
  Interventions: Drug: Arsenic Trioxide
- Without arsenic trioxide therapy (No Intervention): Only receiving cART without arsenic Trioxide after attaining plasma HIV-1 suppression (plasma HIV RNA <50 cp/ml) and CD4+ cell count more than 350 cells/ul over 1 year by cART, without active HCV or HBV infection or opportunistic infections.

INTERVENTIONS:
Drug: Arsenic Trioxide — a arsenic class of mineral, clinically approved for treating acute promyelocytic leukemia
  Other Names: Arsenic Trioxide Injectable Solution
  Arms: Arsenic trioxide combined with cART

SUMMARY:
To evaluate the safety and efficacy of arsenic trioxide combined with cART in eliminating latent HIV-1 reservoir, providing potential strategies for AIDS functional cure.

DETAILED DESCRIPTION:
Although combined antiretroviral therapy (cART) could control human immunodeficiency virus type 1 (HIV-1) infection, the persistence of HIV-1 viral reservoir make it extremely difficult to achieving cure of AIDS. The shock and kill strategy has been extensively practiced. The latency reversing agents (LRAs) could reactivate latent HIV-1 and then the reactivated virus could be eradicated. However, no appropriate activator has been found nor manufactured. Our previous work found that the arsenic trioxide, clinically approved for treating acute promyelocytic leukemia,could efficiently reactivate latent provirus in CD4+T cells from HIV-1 patients and Simian immunodeficiency virus (SIV)-infected macaques, without significant systemic T cell activation and inflammatory responses. In this study, we are going to study the safety of and efficacy of arsenic trioxide combined with cART in 20 HIV-1 infected patients, by observing adverse events,HIV-1 reservoir, HIV-1 load, and some immune index.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection confirmed
2. Receiving HAART more than 12 months.
3. HIV viral-load < 50 copies/ml and CD4+ cell count more than 350 cells/ul.
4. Without serious heart, lung, liver or kidney disease.
5. Participants know about the study and sign informed consent.

Exclusion Criteria:

1. With serious active HBV or HCV infection or opportunistic infections
2. With serious chronic disease such as diabetes, mental illness,et al
3. History of suffering from pancreatitis during HAART.
4. Pregnant or breast-fed.
5. With poor adherence.
6. Unable to complete the follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events of arsenic trioxide combined with cART | 6 Months
  To observe the adverse events of arsenic trioxide combined with cART when treating with HIV-infected patients during the clinical trial

SECONDARY OUTCOMES:
HIV-1 reservoir | 6 Months
  To assay the HIV-1 viral load in the peripheral blood Mono-nuclear cells and plasma

OTHER OUTCOMES:
HIV-specific immunity | 6 Months
  The number of HIV-specific CD4,CD8 and their activity after receiving arsenic trioxide

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Cai, Bachelor, Study Chair — Guangzhou 8th People's Hospital
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu C, Ma X, Liu B, Chen C, Zhang H. HIV-1 functional cure: will the dream come true? BMC Med. 2015 Nov 20;13:284. doi: 10.1186/s12916-015-0517-y. PMID 26588898
- [Background] Chun TW, Engel D, Berrey MM, Shea T, Corey L, Fauci AS. Early establishment of a pool of latently infected, resting CD4(+) T cells during primary HIV-1 infection. Proc Natl Acad Sci U S A. 1998 Jul 21;95(15):8869-73. doi: 10.1073/pnas.95.15.8869. PMID 9671771
- [Background] Deng K, Pertea M, Rongvaux A, Wang L, Durand CM, Ghiaur G, Lai J, McHugh HL, Hao H, Zhang H, Margolick JB, Gurer C, Murphy AJ, Valenzuela DM, Yancopoulos GD, Deeks SG, Strowig T, Kumar P, Siliciano JD, Salzberg SL, Flavell RA, Shan L, Siliciano RF. Broad CTL response is required to clear latent HIV-1 due to dominance of escape mutations. Nature. 2015 Jan 15;517(7534):381-5. doi: 10.1038/nature14053. Epub 2015 Jan 7. PMID 25561180
- [Background] McCoy LE, Weiss RA. Neutralizing antibodies to HIV-1 induced by immunization. J Exp Med. 2013 Feb 11;210(2):209-23. doi: 10.1084/jem.20121827. PMID 23401570
- [Background] Eriksson S, Graf EH, Dahl V, Strain MC, Yukl SA, Lysenko ES, Bosch RJ, Lai J, Chioma S, Emad F, Abdel-Mohsen M, Hoh R, Hecht F, Hunt P, Somsouk M, Wong J, Johnston R, Siliciano RF, Richman DD, O'Doherty U, Palmer S, Deeks SG, Siliciano JD. Comparative analysis of measures of viral reservoirs in HIV-1 eradication studies. PLoS Pathog. 2013 Feb;9(2):e1003174. doi: 10.1371/journal.ppat.1003174. Epub 2013 Feb 14. PMID 23459007
- [Background] Hutter G, Nowak D, Mossner M, Ganepola S, Mussig A, Allers K, Schneider T, Hofmann J, Kucherer C, Blau O, Blau IW, Hofmann WK, Thiel E. Long-term control of HIV by CCR5 Delta32/Delta32 stem-cell transplantation. N Engl J Med. 2009 Feb 12;360(7):692-8. doi: 10.1056/NEJMoa0802905. PMID 19213682
- [Background] Leong YA, Atnerkar A, Yu D. Human Immunodeficiency Virus Playing Hide-and-Seek: Understanding the TFH Cell Reservoir and Proposing Strategies to Overcome the Follicle Sanctuary. Front Immunol. 2017 May 31;8:622. doi: 10.3389/fimmu.2017.00622. eCollection 2017. PMID 28620380
- [Background] Fellmann C, Gowen BG, Lin PC, Doudna JA, Corn JE. Cornerstones of CRISPR-Cas in drug discovery and therapy. Nat Rev Drug Discov. 2017 Feb;16(2):89-100. doi: 10.1038/nrd.2016.238. Epub 2016 Dec 23. PMID 28008168
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Wong JK, Hezareh M, Gunthard HF, Havlir DV, Ignacio CC, Spina CA, Richman DD. Recovery of replication-competent HIV despite prolonged suppression of plasma viremia. Science. 1997 Nov 14;278(5341):1291-5. doi: 10.1126/science.278.5341.1291. PMID 9360926
- [Background] Donahue DA, Wainberg MA. Cellular and molecular mechanisms involved in the establishment of HIV-1 latency. Retrovirology. 2013 Feb 1;10:11. doi: 10.1186/1742-4690-10-11. PMID 23375003
- [Background] Goulder PJ, Watkins DI. HIV and SIV CTL escape: implications for vaccine design. Nat Rev Immunol. 2004 Aug;4(8):630-40. doi: 10.1038/nri1417. No abstract available. PMID 15286729
- [Background] Goonetilleke N, Liu MK, Salazar-Gonzalez JF, Ferrari G, Giorgi E, Ganusov VV, Keele BF, Learn GH, Turnbull EL, Salazar MG, Weinhold KJ, Moore S; CHAVI Clinical Core B; Letvin N, Haynes BF, Cohen MS, Hraber P, Bhattacharya T, Borrow P, Perelson AS, Hahn BH, Shaw GM, Korber BT, McMichael AJ. The first T cell response to transmitted/founder virus contributes to the control of acute viremia in HIV-1 infection. J Exp Med. 2009 Jun 8;206(6):1253-72. doi: 10.1084/jem.20090365. Epub 2009 Jun 1. PMID 19487423
- [Background] Qiao L, Li Y, Xiong G, Liu X, He S, Tong X, Wu S, Hu H, Wang R, Hu H, Chen L, Zhang L, Wu J, Dai F, Lu C, Xiang Z. Effects of altered catecholamine metabolism on pigmentation and physical properties of sclerotized regions in the silkworm melanism mutant. PLoS One. 2012;7(8):e42968. doi: 10.1371/journal.pone.0042968. Epub 2012 Aug 24. PMID 22937004
- [Background] Abaza Y, Kantarjian H, Garcia-Manero G, Estey E, Borthakur G, Jabbour E, Faderl S, O'Brien S, Wierda W, Pierce S, Brandt M, McCue D, Luthra R, Patel K, Kornblau S, Kadia T, Daver N, DiNardo C, Jain N, Verstovsek S, Ferrajoli A, Andreeff M, Konopleva M, Estrov Z, Foudray M, McCue D, Cortes J, Ravandi F. Long-term outcome of acute promyelocytic leukemia treated with all-trans-retinoic acid, arsenic trioxide, and gemtuzumab. Blood. 2017 Mar 9;129(10):1275-1283. doi: 10.1182/blood-2016-09-736686. Epub 2016 Dec 21. PMID 28003274
- [Background] Wang P, Qu X, Wang X, Liu L, Zhu X, Zeng H, Zhu H. As2O3 synergistically reactivate latent HIV-1 by induction of NF-kappaB. Antiviral Res. 2013 Dec;100(3):688-97. doi: 10.1016/j.antiviral.2013.10.010. PMID 24416773